CLINICAL TRIAL: NCT01370499
Title: Long-Term, Open-Label, Safety Study of LY2216684 12 to 18 mg Once Daily as Adjunctive Treatment for Adult Patients With Major Depressive Disorder Who Were Partial Responders to Selective Serotonin Reuptake Inhibitor Treatment
Brief Title: A Study of LY2216684 in Participants With Major Depression Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12849; H9P-JE-LNDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684 + SSRI (Experimental): LY2216684: 12 milligrams (mg) or 18 mg, administered orally, once daily for 52 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  During the open-label phase, all participants started at the 12 mg dose and could have the dose increased to 18 mg after the first week of treatment. During the first 12 weeks, participants were allowed (at scheduled or unscheduled visits) to decrease their dose to 12 mg based on response. After a decrease in dose to 12 mg, participants could have had an increase back up to 18 mg at any scheduled visit based on response and tolerability. After 12 weeks of treatment, participants maintained a stable dose.
  Open-label treatment was followed by a 1-week abrupt discontinuation phase. Participants who either completed study visits through Week 52 or discontinued early from the study for any reason returned 1 week later for follow-up visit. Participants did not receive LY2216684 but continued their SSRI treatment at a stable dose.
  Interventions: Drug: LY2216684; Drug: SSRI

INTERVENTIONS:
Drug: LY2216684
  Other Names: Edivoxetine
Drug: SSRI — Participants were to enter the study taking their current stable SSRI treatment dose and maintain the same dose throughout the study.
  Other Names: Selective Serotonin Reuptake Inhibitor

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of LY2216684 administered once daily in the adjunctive treatment with an Selective Serotonin Reuptake Inhibitors (SSRI) for up to approximately 1 year in participants with Major Depressive Disorder (MDD) who were partial responders to their SSRI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed Study LNBM: NCT01173601 or Study LNBQ: NCT01187407
* Participants must be competent and able to give their own informed consent

Exclusion Criteria:

* Participants that have had or currently have any additional ongoing Diagnostic and Statistical Manual of Mental Disorder, fourth edition, text revision (DSM-IV-TR) Axis I condition other than major depression that was considered the primary diagnosis within 1 year of entering trial
* Participants that have had any anxiety disorder that was considered a primary diagnosis within the past year
* Participants that have a current or previous diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder
* Participants that have a history of substance abuse within the past 1 year, and/or substance dependence within the past 1 year, not including caffeine and nicotine
* Participants that have an Axis II disorder that, in the judgment of the investigator, would interfere with compliance with the study
* Participants that have had a lack of full response of the current depressive episode to 2 or more adequate courses of antidepressant therapy at a clinically appropriate dose for at least 4 weeks, or in the judgment of the investigator, the participant has treatment-resistant depression
* Participants that have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or psychosurgery within the last year
* Participants who are women who are pregnant or breastfeeding
* Participants who, in the opinion of the investigator, are judged to be at serious risk for harm to self or others
* Participants that have a serious or unstable medical illness
* Participants that have any diagnosed medical condition which could be exacerbated by noradrenergic agents
* Participants that have a history of severe allergies to more than 1 class of medication or multiple adverse drug reactions
* Participants that have a history of any seizure disorder (other than febrile seizures)
* Participants that have received treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to entering trial or have a potential need to use an MAOI within 3 days after discontinuation from the study
* Participants that require psychotropic medication other than sedative/hypnotic medication for sleep
* Participants who are taking or have received treatment with any excluded medications within 7 days prior to entering trial
* Participants that have a thyroid stimulating hormone (TSH) level outside the laboratory established reference range. Participants previously diagnosed with hyperthyroidism or hypothyroidism who have been treated with a stable dose of thyroid supplement for at least the past 3 months, and who are clinically and chemically euthyroid will be allowed to participate in the study.
* Participants that have initiated or discontinued hormone therapy within the previous 3 months prior to enrollment
* Participants that have initiated psychotherapy, change in intensity of psychotherapy or other nondrug therapies (such as acupuncture or hypnosis) within 6 weeks prior to enrollment or at any time during the study.
* Participants have a positive urine drug screen (UDS) for any substances of abuse on entering trial
* Participants have significantly violated rules that a participant must comply with during Study LNBM: NCT01173601 or Study LNBQ: NCT01187407

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label study with 1 treatment (12 or 18 milligrams [mg] LY2216684 + SSRI). However, the data were analyzed by the participants' treatment group from 2 parent studies (Study LNBM: NCT01173601 or Study LNBQ: NCT01187407). In these prior, parent studies, participants were randomized to receive Placebo + SSRI or LY2216684 + SSRI.
Groups:
- LY2216684 + SSRI (Placebo Prior Study): LY2216684: 12 mg or 18 mg, administered orally, once daily for 52 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- LY2216684 + SSRI (LY2216684 Prior Study): LY2216684: 12 mg or 18 mg, administered orally, once daily for 52 weeks, adjunctive to an SSRI
Period: Overall Study
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Started | 195 | 93
Entered Abrupt Discontinuation Phase | 188 | 85 (One participant who entered the abrupt discontinuation phase did not receive study drug.)
Received at Least 1 Dose of Study Drug | 195 | 92
Completed | 84 | 49
Not Completed | 111 | 44
Not completed — Adverse Event | 38 | 12
Not completed — Lack of Efficacy | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Sponsor Decision | 41 | 15

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- LY2216684 + SSRI (Placebo Prior Study); LY2216684 + SSRI (LY2216684 Prior Study): LY2216684: 12 mg or 18 mg, administered orally, once daily for 52 weeks, adjunctive to an SSRI
- Total: Total of all reporting groups
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study) | Total
Number analyzed (Participants) | 195 | 93 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.28 (9.41) | 37.40 (9.18) | 38.68 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 45 | 133
  Male | 107 | 48 | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 195 | 93 | 288
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 195 | 93 | 288

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Events
Description: Clinically significant events were defined as serious adverse events, regardless of causality. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through 52 weeks
Population: All participants who took at least one dose of study medication and did not discontinue from the study for the reason 'Lost to follow-up' at the first post-baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 195 | 92
Participants
  Contusion | 0 | 1
  Hyperglycaemia | 0 | 1
  Subdural hygroma | 1 | 0

2. Secondary Outcome: Percentage of Participants With Suicidal Behaviors and Ideations Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation was defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which included a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as treatment-emergent (TE) if not present at baseline. Percentage of participants was calculated by dividing the number of participants with suicide-related events by the total number of participants at risk, multiplied by 100%. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through 52 weeks
Population: All participants who took at least one dose of study medication and had a baseline and at least one post-baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 195 | 92
percentage of participants
  TE of suicidal ideation | 8.72 | 8.70
  Suicidal behavior | 0.51 | 0.00

3. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score and Individual Items
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items are rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 195 | 93
units on a scale
  MADRS total score | -4.33 (0.69) | -6.63 (1.00)
  Apparent sadness | -0.36 (0.10) | -1.01 (0.16)
  Reported sadness | -0.51 (0.12) | -0.92 (0.20)
  Inner tension | -0.53 (0.10) | -0.85 (0.18)
  Reduced sleep | -0.49 (0.12) | -0.33 (0.19)
  Reduced appetite | -0.24 (0.08) | -0.25 (0.16)
  Concentration difficulties | -0.72 (0.11) | -1.12 (0.17)
  Lassitude | -0.71 (0.09) | -0.78 (0.16)
  Inability to feel | -0.41 (0.11) | -0.77 (0.14)
  Pessimistic thoughts | -0.31 (0.09) | -0.63 (0.14)
  Suicidal thoughts | -0.19 (0.06) | -0.25 (0.07)

4. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Clinical Global Impression - Severity (CGI-S)
Description: Clinical Global Impression - Severity (CGI-S) measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 195 | 93
units on a scale | -0.80 (0.10) | -0.78 (0.13)

5. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Fatigue Associated With Depression (FAsD) Average Score and Subscale Scores
Description: The FAsD is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The "Experience Score" was derived by taking the mean of Items 1 through 6, the "Impact Score" was derived by taking the mean of Items 7 through 13 (applicable items only), and the "Average Score" was the mean of Items 1 through 13 (derived by taking the mean of all applicable items for each participant). Item 12 applied only to participants with a spouse or significant other and Item 13 applied to participants who had a job or who went to school. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 183 | 86
units on a scale
  Average score | -0.32 (0.07) | -0.18 (0.08)
  Experience score | -0.28 (0.08) | -0.15 (0.09)
  Impact score | -0.34 (0.07) | -0.19 (0.08)

6. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Hospital Anxiety and Depression Scale (HADS) Depression and Anxiety Subscale Scores
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. The anxiety subscale score is the sum of the 7 odd-numbered items and depression subscale score is the sum of the 7 even-numbered items, giving maximum scores of 21 for each subscale. Scores of 11 or more on either subscale were considered to be a 'significant' case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal'. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 189 | 87
units on a scale
  Anxiety | -1.46 (0.28) | -0.55 (0.38)
  Depression | -1.95 (0.34) | -1.24 (0.44)

7. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Sheehan Disability Scale (SDS) Total Score and Subscale Scores
Description: The SDS Global Functional Impairment Score (total score) and subscores were completed by the participant and were used to assess the effect of the participant's symptoms on his or her work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. The Global Functional Impairment Score is the sum of the 3 items, and scores ranged from 0 to 30 with high values indicating greater disruption in the participant's work life (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 177 | 81
units on a scale
  Global functional impairment score: number analyzed (Participants) | 117 | 81
  Global functional impairment score | -3.11 (0.63) | -2.37 (0.70)
  Work impairment score: number analyzed (Participants) | 131 | 58
  Work impairment score | -0.98 (0.29) | -1.42 (0.42)
  Social life impairment score | -1.01 (0.21) | -0.66 (0.25)
  Family life impairment score | -1.10 (0.20) | -0.55 (0.24)

8. Secondary Outcome: Change From Baseline to 52 Week Endpoint in EuroQol Questionnaire - 5 Dimension (EQ-5D)
Description: The 5Q-5D Visual Analog Scale is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score is self-reported using a visual analogue scale, marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 177 | 81
units on a scale | 9.445 (1.846) | 9.989 (2.288)

9. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is a self-administered 16-item questionnaire measuring degree of enjoyment and satisfaction experienced in various areas of daily life during the past week on a 5-point Likert scale (1=very poor and 5=very good). The total possible scores range from 16 to 80. Higher scores indicate higher levels of enjoyment/satisfaction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All enrolled participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 177 | 81
units on a scale | 6.28 (1.30) | 5.19 (1.58)

10. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The CPFQ is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item is scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total scores ranged from 7 to 42. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All participants who took at least one dose of study medication and had a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 183 | 86
units on a scale | -4.02 (0.54) | -2.53 (0.75)

11. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Arizona Sexual Experiences (ASEX) Scale
Description: The Arizona Sexual Experiences (ASEX) scale is used to assess sexual functioning in both males and females. The ASEX total score for the male and female version is calculated as the sum of the responses (rated from 1 [extremely] to 6 [no/never]) to the 5 items of the ASEX scale. Total scores ranged from 5 to 30, with higher scores indicating greater sexual dysfunction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All participants who took at least one dose of study medication and had a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 183 | 85
units on a scale | -0.65 (0.39) | -0.40 (0.55)

12. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Blood Pressure
Description: Blood pressure measurements were collected when the participant was in a sitting position. Three measurements of sitting blood pressure collected at approximately 1-minute intervals at every visit were averaged and used as the value for the visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All participants who took at least one dose of study medication and had a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 195 | 92
millimeters of mercury (mmHg)
  Sitting systolic blood pressure | 6.66 (0.93) | 3.68 (1.28)
  Sitting diastolic blood pressure | 7.55 (0.83) | 6.34 (1.03)

13. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Pulse Rate
Description: Pulse measurements were collected when the participant was in a sitting position. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for pooled investigative site and visit, baseline score, and baseline score-by-visit interaction.
Time Frame: Baseline, 52 weeks
Population: All participants who took at least one dose of study medication and had a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study)
Number analyzed (Participants) | 195 | 92
beats per minute (bpm) | 17.00 (1.24) | 10.98 (1.49)

ADVERSE EVENTS:
Groups:
- LY2216684 + SSRI (Placebo Prior Study); LY2216684 + SSRI (LY2216684 Prior Study): LY2216684: 12 mg or 18 mg, administered orally, once daily for 52 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes all randomized participants who received at least 1 dose of study drug.
- LY2216684 + SSRI (Placebo Prior Study) DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all randomized participants who received at least 1 dose of study drug and abruptly discontinued LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- LY2216684 + SSRI (LY2216684 Prior Study) DC Phase: No study drug was administered. Participants were to maintain their SSRI treatment at a stable dose for 1 week.
  Includes all participants who received at least 1 dose of study drug and abruptly discontinued LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
Arm/Group | LY2216684 + SSRI (Placebo Prior Study) | LY2216684 + SSRI (LY2216684 Prior Study) | LY2216684 + SSRI (Placebo Prior Study) DC Phase | LY2216684 + SSRI (LY2216684 Prior Study) DC Phase
Serious Adverse Events (participants affected / at risk) | 1/195 | 2/92 | 0/188 | 0/84
Other Adverse Events (participants affected / at risk) | 158/195 | 67/92 | 9/188 | 3/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 + SSRI (Placebo Prior Study) (N=195) | LY2216684 + SSRI (LY2216684 Prior Study) (N=92) | LY2216684 + SSRI (Placebo Prior Study) DC Phase (N=188) | LY2216684 + SSRI (LY2216684 Prior Study) DC Phase (N=84)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 + SSRI (Placebo Prior Study) (N=195) | LY2216684 + SSRI (LY2216684 Prior Study) (N=92) | LY2216684 + SSRI (Placebo Prior Study) DC Phase (N=188) | LY2216684 + SSRI (LY2216684 Prior Study) DC Phase (N=84)
Palpitations (Cardiac disorders) | 36 (38) | 12 (12) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 62 (77) | 17 (20) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 19 (20) | 7 (7) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 26 (29) | 8 (10) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (14) | 3 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 56 (94) | 29 (39) | 3 (3) | 0 (0)
Blood pressure increased (Investigations) | 11 (11) | 0 (0) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 25 (31) | 7 (11) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 21 (28) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 17 (45) | 7 (8) | 2 (2) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 14 (14) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 10 (10) | 4 (4) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 33 (33) | 16 (16) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days